CLINICAL TRIAL: NCT06929741
Title: Cross-cultural Adaptation and Validation of a Turkish Version of the Arthritis Self-Efficacy Scale-8 (ASES-8) for Patients With Knee Osteoarthritis
Brief Title: Turkish Version of the Arthritis Self-Efficacy Scale-8
Acronym: T-ASES-8
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/211
Record Dates: First submitted 2025-04-07; First posted 2025-04-16 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Knee Osteoarthristis; Self Efficacy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Knee Osteoarthritis (KOA)

SUMMARY:
Self-efficacy is a psychosocial construct that reflects an individual's confidence in their ability to perform specific tasks, focusing more on one's belief in their abilities than on actual performance. This concept is especially important in knee osteoarthritis (KOA) management, as it can significantly influence overall health and treatment outcomes, and it is considered a modifiable trait.

KOA is one of the most common musculoskeletal disorders worldwide, substantially impacting quality of life due to symptoms such as limited mobility, chronic pain, and joint stiffness. These symptoms can hinder daily activities and potentially lead to social isolation. In patients with KOA, a strong sense of self-efficacy can improve symptom management and increase participation in physical activities. Research indicates that patients with higher self-efficacy are more likely to engage actively in rehabilitation programs and achieve their treatment goals. Consequently, various self-efficacy measurement tools have been developed to better understand patients' perceptions of their condition and the extent of their disability, which in turn aids in formulating strategies to enhance self-efficacy and optimize treatment responses.

The Arthritis Self-Efficacy Scale (ASES) is widely used to assess self-efficacy in managing pain, physical functions, and other symptoms associated with arthritis. Compared to other self-efficacy instruments, the ASES has a longstanding history and is particularly applicable to KOA. Its validity and reliability have been confirmed through several studies. Initially developed as a 20-item scale with three subscales evaluating physical function, pain, and other symptoms, a shorter version-the eight-item ASES-8-was later created. This abbreviated version includes two items from the pain subscale, four items from the other symptoms subscale, and two additional items addressing fatigue and pain prevention during daily activities. Each item is rated on a scale from 1 (very uncertain) to 10 (very certain), indicating the patient's level of confidence in managing their condition.

Although the ASES-8 has been validated in several languages, it has not yet been translated into Turkish or culturally adapted for Turkish patients with KOA. Cross-cultural adaptation of patient-reported outcome measures (PROMs) requires rigorous methodologies to ensure both accurate translation and the preservation of content validity. Reliable, valid, and culturally sensitive instruments are essential for developing effective interventions for Turkish-speaking patients with KOA. Therefore, this study aims to translate and cross-culturally adapt the ASES-8 into Turkish and evaluate the reliability and validity of the resulting instrument.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of knee osteoarthritis (KOA) according to the American College of Rheumatology (ACR) criteria
* Sufficient language skills to understand and complete the scale
* Provision of informed consent

Exclusion Criteria:

* Health conditions unsuitable for a self-management program
* Behavioral or cognitive issues that could hinder the assessment process
* Unstable angina or uncontrolled heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study targets adult patients aged 18 years and older who have been diagnosed with knee osteoarthritis (KOA) based on the American College of Rheumatology (ACR) criteria. Participants must possess sufficient language proficiency to understand and complete the Turkish version of the ASES-8 scale and must be willing to provide informed consent. The study excludes individuals with health conditions that render them unsuitable for self-management programs, those with behavioral or cognitive impairments that could interfere with the assessment process, and patients with unstable angina or uncontrolled heart failure.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Construct Validity and Reliability of the Turkish ASES-8 | 1 month
  Self-Efficacy in Knee Osteoarthritis (KOA) Management
  The primary outcome of our study is to assess the level of self-efficacy in managing KOA among Turkish-speaking patients. This is operationalized through the culturally adapted version of the Arthritis Self-Efficacy Scale-8 item version (ASES-8).
  Key Features of the Primary Outcome Measure:
  Instrument Overview:
  The ASES-8 is designed to evaluate the patient's confidence in managing key symptoms associated with KOA-including pain, functional limitations, fatigue, and pain prevention during daily activities. Unlike performance-based tests, this instrument focuses on patients' beliefs about their own abilities to manage these aspects, which is crucial for effective self-management.
  Measurement Details:
  Item Structure: The ASES-8 consists of eight items. Two items are derived from the pain subscale, four from the other symptoms subscale, and two additional items address fatigue and preventive strategies against pain during daily ac

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided